CLINICAL TRIAL: NCT02773823
Title: A Comprehensive Intervention Study on Klotho Gene Methylation and Cardiovascular Risk Factors
Brief Title: A Behavior Intervention Study on Cardiovascular Health Among Chinese Obese Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Qiqiang He, Professor, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81372973
Record Dates: First submitted 2016-05-07; First posted 2016-05-16 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases
Keywords: obesity; children; cardiovascular health; intervention study
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Lifestyle intervention includes diet instruction and exercise intervention:
  1. Diet instruction: The children were asked to increase fruit/vegetables consumption, reduce high fat food, etc.
  2. Exercise intervention: The children participated sports 60 min/day,5d/week for 8 months.
  Interventions: Behavioral: Intervention group
- Control (No Intervention): No intervention in the group with "control".

INTERVENTIONS:
Behavioral: Intervention group — Diet instruction for 3-4 times/semester,exercise 60min/day for 5d/week for 8 months.
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the effects of comprehensive behavior on cardiovascular health among obese schoolchildren. The intervention methods include dietary instruction and exercise intervention. The main outcomes are weight, body mass index, blood pressure, lipids and glucose.

DETAILED DESCRIPTION:
Two public primary schools of a similar size were selected. They were allocated either to the intervention or control group. Children in Grade 4th and 5th in each school were invited to participate in the physical examination (height and weight measures).Obese children based on Chinese BMI cut-off points were included in this study.Children in the intervention group were encouraged to take healthy diet habits and increased their physical activity.After eight months healthy behavior intervention, Children's height, weight, waist, hip, blood pressure, cardiorespiratory fitness will be measured. Fasting blood will be taken to measure lipids and glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Obese children; Aged 8-12 years old.

Exclusion Criteria:

* History of cardiovascular diseases and diabetes; Disability.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Body weight of study children | 8 months
  Body weight will be measured with light clothes using a scale to the nearest 0.1 kg.
Body mass index of study children | 8 months
  Body mass index is defined as the individual's body weight divided by the square of his or her height (height is measured using a non- stretchable tape suspended from the wall is recorded to the nearest 0.1 cm).
Waist circumference of study children | 8 months
  Waist circumference will be measured using a tape around his or her bare abdomen to the nearest 0.1 cm.
Blood pressure | 8 months
  Blood pressure will be measured three times by auscultation method with appropriate cuff size after 20 minutes of rest.The average of the blood pressure measurements is defined as hypertension if it was >95th percentile according to their age, gender and height percentile.
Blood lipids | 8 months
  Blood samples will be obtained in the morning by venipuncture after an overnight fast. Serum lipid profiles (total cholesterol ,triglycerides, low-density lipoprotein, high-density lipoprotein) will be measured using routine enzymatic methods.
Blood glucose | 8 months
  Blood samples is obtained in the morning by venipuncture after an overnight fast. The glucose oxidase method was used in the determination of blood glucose levels.
cardiorespiratory fitness of study children | 8 months
  Cardiorespiratory refers to the ability of the circulatory and respiratory systems to supply oxygen to skeletal muscles during sustained physical activity. It is measured by 20 meter shuttle-run test.

SECONDARY OUTCOMES:
Well-being of study children | 8 months
  Well-being will be measured by The WHO 5-item Well-Being Index (WHO-5), which is a short screening instrument for the detection of depression in the general population,
Depression of study children | 8 months
  The Depression Self-Rating Scale for Children (DSRSC) will be used for screening depression in children.

CONTACTS AND LOCATIONS:
Overall Officials: Qiqiang He, PhD, Principal Investigator — Wuhan University
Locations (1):
- Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hu FB, Manson JE, Stampfer MJ, Colditz G, Liu S, Solomon CG, Willett WC. Diet, lifestyle, and the risk of type 2 diabetes mellitus in women. N Engl J Med. 2001 Sep 13;345(11):790-7. doi: 10.1056/NEJMoa010492. PMID 11556298
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] He QQ, Wong TW, Du L, Jiang ZQ, Yu TS, Qiu H, Gao Y, Liu WJ, Wu JG. Physical activity, cardiorespiratory fitness, and obesity among Chinese children. Prev Med. 2011 Feb;52(2):109-13. doi: 10.1016/j.ypmed.2010.11.005. Epub 2010 Nov 23. PMID 21108961
- [Background] Semba RD, Cappola AR, Sun K, Bandinelli S, Dalal M, Crasto C, Guralnik JM, Ferrucci L. Plasma klotho and cardiovascular disease in adults. J Am Geriatr Soc. 2011 Sep;59(9):1596-601. doi: 10.1111/j.1532-5415.2011.03558.x. Epub 2011 Aug 24. PMID 21883107
- [Background] Thompson D, Markovitch D, Betts JA, Mazzatti D, Turner J, Tyrrell RM. Time course of changes in inflammatory markers during a 6-mo exercise intervention in sedentary middle-aged men: a randomized-controlled trial. J Appl Physiol (1985). 2010 Apr;108(4):769-79. doi: 10.1152/japplphysiol.00822.2009. PMID 20368384